CLINICAL TRIAL: NCT01484652
Title: A Phase 3 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Evaluation of the Safety and Analgesic Efficacy of COV795 in Moderate to Severe Post-Operative Bunionectomy Pain Followed by an Open-Label Extension
Brief Title: Safety and Efficacy of COV795 in Moderate to Severe Post-Operative Bunionectomy Pain With an Open-label Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COV15000182
Record Dates: First submitted 2011-11-28; First posted 2011-12-02 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Pain, Postoperative; Bunion
Keywords: Moderate Post-Operative Pain; Severe Post-Operative Pain; Bunionectomy
MeSH Terms: conditions — Pain, Postoperative; Bunion | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- COV795 (Experimental)
  Interventions: Drug: COV795
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COV795 — 2 tablets taken every 12 hours
  Other Names: MNK795
  Arms: COV795
Drug: Placebo — 2 tablets taken every 12 hours
  Arms: Placebo

SUMMARY:
The primary objective of this study is to show the effectiveness of repeated doses of COV795 versus placebo, using the summed pain intensity difference over the first 48 hours in subjects with acute moderate to severe pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria

1. Complete the informed consent process as documented by signed informed consent form(s).
2. Be in generally good health.
3. Be 18 to 75 years of age, inclusively at the time of screening.
4. Be scheduled for a primary unilateral first metatarsal bunionectomy (with no collateral procedures).
5. Have a body mass index ≤33 kg/m2.
6. Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant for the duration of the study, surgically sterile or at least two years postmenopausal, or practicing an acceptable form of birth control for at least 2 months
7. Male subjects must be sterile or commit to the use of a reliable method of birth control
8. Be classified as Physical status 1 (PS-1) to PS-2 by the American Society of Anesthetists (ASA) Physical Status Classification System.
9. Be willing to complete the pain evaluations and return to the clinic as scheduled.

Exclusion Criteria

1. Have an uncontrolled medical condition, serious intercurrent illness, clinically significant general health condition, or extenuating circumstance that may significantly decrease study compliance or otherwise preclude their participation in the study.
2. Have a clinically significant abnormal electrocardiogram (ECG) at screening
3. Have had any type of gastric bypass surgery or have a gastric band.
4. Have previous abdominal surgery within the past year or history of abdominal adhesions, known or suspected paralytic ileus.
5. Have a history of any medical condition that would alter the absorption, distribution, metabolism or excretion of COV795
6. Have a history of severe bronchial asthma, hypercarbia, or hypoxia
7. Have a clinically significant abnormality on their clinical laboratory values
8. Have Addison's disease, benign prostatic hyperplasia, or kidney disease
9. Have donated blood or blood components within 3 months prior to the screening visit.
10. Have a known allergy or hypersensitivity to any opioid analgesics, anesthetics, acetaminophen, Non-steroid anti-inflammatory drugs (NSAIDs).
11. Have a history of intolerance to short term opioid use.
12. Unwilling to discontinue certain prohibited medications within the allotted time before surgery and throughout the duration of the study. Have taken certain drugs within the indicated times before surgery.
13. Have a history of substance or alcohol abuse and/or a positive result on drug screening.
14. Have a positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at the screening visit.
15. Have dysphagia and/or cannot swallow study medication whole.
16. Have a history of migraine or frequent headaches, seizures, or are currently taking anticonvulsants.
17. Have previously participated in a clinical trial using COV795 or had a bunionectomy in the last 3 months.
18. Received any investigational drugs or devices within 4 weeks prior to the screening visit.
19. Other criteria as specified in the trial protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Trovare Clinical Research, Inc., Bakersfield, California
  - Lotus Clinical Research, LLC, Pasadena, California
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Jean Brown Research, Inc., Salt Lake City, Utah

REFERENCES:
- [Derived] Singla N, Barrett T, Sisk L, Kostenbader K, Young J. Assessment of the safety and efficacy of extended-release oxycodone/acetaminophen, for 14 days postsurgery. Curr Med Res Opin. 2014 Dec;30(12):2571-8. doi: 10.1185/03007995.2014.957824. Epub 2014 Oct 13. PMID 25157951
- [Derived] Singla N, Barrett T, Sisk L, Kostenbader K, Young J, Giuliani M. A randomized, double-blind, placebo-controlled study of the efficacy and safety of MNK-795, a dual-layer, biphasic, immediate-release and extended-release combination analgesic for acute pain. Curr Med Res Opin. 2014 Mar;30(3):349-59. doi: 10.1185/03007995.2013.876979. Epub 2014 Jan 10. PMID 24351079

RESULTS

PARTICIPANT FLOW:
Groups:
- COV795; Placebo: 2 tablets taken every 12 hours at Hour 0, 12, 24, and 36; total of 4 doses
Period: Overall Study
Arm/Group | COV795 | Placebo
Started | 166 | 163
Completed | 151 | 142
Not Completed | 15 | 21

BASELINE CHARACTERISTICS:
Population: The analysis population for baseline characteristics includes all 329 subjects who received at least one dose of study treatment. The subjects were assigned 2 cohort classifications. Cohort 1 included 26 subjects enrolled under the original protocol and amendment 1. Cohort 2 is the remainder of the 303 subjects enrolled after amendment 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | COV795 | Placebo | Total
Number analyzed (Participants) | 166 | 163 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.17) | 44.6 (14.14) | 43.4 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 135 | 280
  Male | 21 | 28 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 51 | 47 | 98
  White | 98 | 103 | 201
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 44 | 82
  Not Hispanic or Latino | 128 | 119 | 247
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SPID48 (Summed Pain Intensity Difference)
Description: Pain intensity (PI) is measured using the 11-point (0-10) Numeric Pain Rating Scale (NPRS) score. PID is the arithmetic difference in NPRS score at the time point of interest from the baseline score. SPID48 is the sum of time-weighted PID scores measured 22 times over the 48 hour assessment period, with a total score ranging from -480 (worst) to 480 (best). A higher SPID value indicates greater pain relief.
Time Frame: 48 hours
Population: The analysis population for the primary outcome measure was the modified intent-to-treat population (mITT). The mITT analysis population includes 303 subjects from Cohort 2. Missing pain intensity difference scores were imputed using a multiple imputation method.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | COV795 | Placebo
Number analyzed (Participants) | 150 | 153
scores on a scale | 114.9 (7.64) | 66.9 (7.6)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) span the entire study, ie, the double-blind and open-label extension phases. Other Adverse Events reflects data from the double-blind phase of the study.
Description: Subjects who received at least one dose of COV795 during the double-blind phase or open-label phase are included in the SAE COV795 group summary. Subjects who only received placebo during the entire study are included in the Placebo group summary.
Arm/Group | COV795 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/235 | 1/94
Other Adverse Events (participants affected / at risk) | 89/166 | 35/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COV795 (N=235) | Placebo (N=94)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Pregnancy test urine positive (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | COV795 (N=166) | Placebo (N=163)
Constipation (Gastrointestinal disorders) | 7 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 51 | 9
Vomiting (Gastrointestinal disorders) | 15 | 0
Edema peripheral (General disorders) | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Dizziness (Nervous system disorders) | 22 | 2
Headache (Nervous system disorders) | 16 | 8
Hypoaesthesia (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 6 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Hot flush (Vascular disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No